CLINICAL TRIAL: NCT04218201
Title: Subthreshold Opioid Use Disorder Prevention (STOP) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-00535
Record Dates: First submitted 2019-12-23; First posted 2020-01-06 (Actual); Results first posted 2025-02-21 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Opioid-use Disorder
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subthreshold Opioid Use Disorder Prevention(STOP) Intervention (Experimental): At baseline, patient participants in the STOP arm will receive the intervention components of brief advice from their PCP and a video doctor , printed educational materials, interaction with the NCM, and telephone health coaching. Brief advice will be delivered by the patient participant's PCP as part of the medical visit or via phone call. Before the encounter with the patient participant, PCPs will receive a brief printed summary report from the research staff. During the baseline visit, patient participants also meet with the research staff to view a video on tablet or desktop computer that reinforces the PCP's counseling.
  Interventions: Behavioral: PCP brief advice; Behavioral: Video doctor; Behavioral: Telephone health coaching; Behavioral: Nurse Care Manager (NCM) intervention
- Enhanced Usual Care (EUC) (No Intervention): PCPs will conduct primary care as usual, without the support of the NCM. At the baseline visit, patient participants receive an educational pamphlet and view a short video on overdose and cancer screening. The pamphlet includes information about preventing opioid-related overdose, including how to obtain a naloxone kit. The video content will feature the health benefits of exercise. It will be viewed on a tablet or desktop computer and will be approximately 2 minutes long. All EUC patient participants receive the same video, which is not tailored to the responses given on their questionnaires. There is no study intervention after the baseline visit.

INTERVENTIONS:
Behavioral: PCP brief advice — Brief advice will be delivered by the patient participant's PCP as part of the medical visit or via phone call. Before the encounter with the patient participant, PCPs will receive a brief printed summary report from the research staff. The summary advises the PCP that their patient participant screened positive for risky opioid use, lists the patient participant's screening results (TAPS Tool +/- COMM) and gives a suggested counseling script. The counseling script will include specific advice on opioid-related risks, will inform patient participants of resources to help them reduce their risk, and will include a recommendation to reduce their risk behavior.
  Arms: Subthreshold Opioid Use Disorder Prevention(STOP) Intervention
Behavioral: Video doctor — During the baseline visit with the research staff, patient participants will view a video on tablet or desktop computer that reinforces the PCP's counseling. The video is a recording of a provider delivering brief advice about opioid use that includes the same elements covered in the summary report outlined above.
  Arms: Subthreshold Opioid Use Disorder Prevention(STOP) Intervention
Behavioral: Telephone health coaching — All patient participants in the STOP arm will receive telephonic health coaching sessions at approximately 2- and 4-weeks post-baseline. Patient participants who may benefit from additional coaching (for example, those who do not improve or who experience clinical worsening of unhealthy opioid use) may receive additional coaching sessions (approximately 4 sessions) from the telephone health coach. Coaching is delivered from a centralized call center, by staff that receive standardized training and supervision. To the extent possible, calls will be scheduled at the patient participant's convenience (e.g., evenings, weekends).
  Arms: Subthreshold Opioid Use Disorder Prevention(STOP) Intervention
Behavioral: Nurse Care Manager (NCM) intervention — NCMs will provide health education and counseling on risk reduction, overdose prevention and self-management skills. Patient participants will be asked to participate in a baseline visit with the NCM, which will occur on the same day as the baseline research visit if possible. The NCM continues working with patients in the STOP condition throughout their 12 months of study participation. Following the initial visit with the NCM, the frequency of visits depends on patient participant needs.
  Arms: Subthreshold Opioid Use Disorder Prevention(STOP) Intervention

SUMMARY:
The Subthreshold Opioid Use Disorder Prevention (STOP) trial will test the efficacy of a primary care intervention to reduce opioid use and overdose risk, and prevent progression to OUD, in adults with unhealthy use of illicit or prescribed opioids. STOP is a collaborative care model. A cluster-randomized trial, conducted in 5 primary care sites, with 100 PCPs and 300adult primary care patients, will test the efficacy of STOP versus enhanced usual care (EUC). The STOP intervention, if proven efficacious, will provide a solution to preventing OUD among patients who are most at risk, thus addressing a key aspect of the current opioid crisis.

DETAILED DESCRIPTION:
This cluster randomized trial, conducted in primary care clinics and randomized at the level of the PCP, will compare the STOP intervention to enhanced usual care (EUC) for 12 months. Patients who are eligible and enroll will receive the intervention according to the assignment of their PCP. In the EUC arm, PCPs conduct primary care as usual, without support of the nurse care manager. Patient participants receive an educational pamphlet about overdose prevention and watch a brief video on "healthy living" that is not specific to substance use. In the STOP arm, PCPs and their enrolled patient participants receive the STOP intervention, consisting of a NCM, brief advice about health risks of opioid misuse, and telephone health coaching. Patient participants in either arm who are found by clinical providers to have developed a moderate-severe OUD at any time during the study can be offered medication for OUD and linked to treatment by clinical staff in the EUC arm, and the NCM in the STOP arm, to formal assessment and MOUD treatment.

ELIGIBILITY:
PCP Inclusion Criteria

* Licensed medical professional (MD, DO, PA, NP).
* Currently providing care to approximately 4 or more adult patients (18 years or older) who are receiving chronic opioid treatment and/or have risky opioid use.
* Total patient volume is approximately 40 or more adult patients (18 years or older) per week on a typical week
* Willing to be randomized to either of the two study conditions

Patient Participant Inclusion Criteria

* PCP is enrolled in the study.
* Age 18 years or older at time of prescreening.
* Proficient in spoken and written English, as determined by patient self-report and research staff evaluation.
* Risky opioid use in the past 90 days from date of prescreening, as determined by a TAPS score >1 for heroin and/or prescription opioids and/or a positive response (>Never) to any of the three COMM items indicating taking more opioid medication than prescribed
* Access to phone that can receive text messages, and access to internet (via smartphone, tablet, or computer), per patient self-report.
* Able to provide informed consent.

PCP Exclusion Criteria:

* Planning to resign from the clinic in the next 24 months, per PCP self-report.
* Planning to change their schedule in the next 24 months such that they would no longer meet the inclusion criteria for patient volume, per PCP self-report.

Patient Participant Exclusion Criteria:

* Patients with moderate-severe OUD, defined as meeting 4 or more DSM-5 criteria for OUD at screening, as assessed by research staff using the modified-CIDI opioid items.
* Receiving MOUD or engaged in an opioid treatment program in the past 30 days from screening date, per patient self-report.
* Receiving opioids for end of life care, per patient self-report.
* Pregnancy (females age 18-50), as determined by patient self-report at the time of screening.
* Are currently in jail, prison, or other overnight facility as required by court of law or have pending legal action that could prevent participation in study activities.
* Plan to leave the area or the clinical practice within the next 12 months, per patient self-report.
* Other factors that may cause harm or increased risk to the participant or close contacts or preclude the patient's full adherence with or completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2024-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer McNeely, MD, Principal Investigator — NYU Langone
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification, with permission from the lead investigator.
Supporting Information: Study Protocol, SAP
Time Frame: Data sets for CTN protocols will be available after (1) the primary paper has been accepted for publication, or (2) the data is locked for more than 18 months, whichever comes first
Access Criteria: Anyone who wishes to access the data. Any purpose. Data are available indefinitely at (https://datashare.nida.nih.gov/).

REFERENCES:
- [Derived] Rostam-Abadi Y, Liebschutz JM, Subramaniam G, Stone R, Appleton N, Mazel S, Alexander K, Brill SB, Case A, Gelberg L, Gordon AJ, Hong H, Incze MA, Kawasaki SS, Kim T, Kline M, Lovejoy TI, McCormack J, Zhang S, McNeely J. Understanding the characteristics and comorbidities of primary care patients with risky opioid use: Baseline data from the multi-site "Subthreshold Opioid Use Disorder Prevention" (STOP) Trial. J Gen Intern Med. 2025 Sep;40(12):2906-2915. doi: 10.1007/s11606-025-09613-4. Epub 2025 Jun 2. PMID 40457116
- [Derived] Liebschutz JM, Subramaniam GA, Stone R, Appleton N, Gelberg L, Lovejoy TI, Bunting AM, Cleland CM, Lasser KE, Beers D, Abrams C, McCormack J, Potter GE, Case A, Revoredo L, Jelstrom EM, Kline MM, Wu LT, McNeely J. Subthreshold opioid use disorder prevention (STOP) trial: a cluster randomized clinical trial: study design and methods. Addict Sci Clin Pract. 2023 Nov 18;18(1):70. doi: 10.1186/s13722-023-00424-8. PMID 37980494

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Randomization occurred at the level of the PCP. Patients who were eligible and enrolled received the intervention according to the assignment of their PCP.
Groups:
- Subthreshold Opioid Use Disorder Prevention(STOP) Intervention - Patients: At baseline, patient participants in the STOP arm will receive the intervention components of brief advice from their PCP and a video doctor , printed educational materials, interaction with the NCM, and telephone health coaching. Brief advice will be delivered by the patient participant's PCP as part of the medical visit or via phone call. Before the encounter with the patient participant, PCPs will receive a brief printed summary report from the research staff. During the baseline visit, patient participants also meet with the research staff to view a video on tablet or desktop computer that reinforces the PCP's counseling.
- STOP Intervention - Primary Care Providers (PCPs): PCPs of participants in the STOP Intervention arm.
- Enhanced Usual Care (EUC) - Patients: PCPs will conduct primary care as usual, without the support of the NCM. At the baseline visit, patient participants receive an educational pamphlet and view a short video on overdose and cancer screening. The pamphlet includes information about preventing opioid-related overdose, including how to obtain a naloxone kit. The video content will feature the health benefits of exercise. It will be viewed on a tablet or desktop computer and will be approximately 2 minutes long. All EUC patient participants receive the same video, which is not tailored to the responses given on their questionnaires. There is no study intervention after the baseline visit.
- EUC - PCPs: PCPs of participants in the EUC arm.
Period: Overall Study
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention - Patients | STOP Intervention - Primary Care Providers (PCPs) | Enhanced Usual Care (EUC) - Patients | EUC - PCPs
Started | 88 | 58 | 114 | 61
Completed | 79 | 49 | 109 | 55
Not Completed | 9 | 9 | 5 | 6
Not completed — Death | 0 | 0 | 2 | 0
Not completed — Unable to contact participant | 4 | 0 | 3 | 0
Not completed — Practical problems (e.g., no childcare or transportation) | 3 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0
Not completed — PCP plans to leave practice | 0 | 8 | 0 | 5
Not completed — Reduced panel | 0 | 0 | 0 | 1
Not completed — No longer interested in participating | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Subthreshold Opioid Use Disorder Prevention(STOP) Intervention - PCPs: PCPs of participants in the STOP arm.
- Enhanced Usual Care (EUC) - PCPs: PCPs of participants in the EUC arm.
- Total: Total of all reporting groups
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention - Patients | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention - PCPs | Enhanced Usual Care (EUC) - Patients | Enhanced Usual Care (EUC) - PCPs | Total
Number analyzed (Participants) | 88 | 58 | 114 | 60 | 320
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.1 (13.31) | 41.4 (7.6) | 56.9 (12.09) | 43.3 (12.23) | 55.7 (12.68)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 23 | 16 | 51 | 26 | 116
  Female | 65 | 38 | 63 | 34 | 200
  Unknown or Not Reported | 0 | 4 | 0 | 0 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 8 | 0 | 13 | 22
  Native Hawaiian or Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 21 | 1 | 22 | 1 | 45
  White | 60 | 38 | 83 | 41 | 222
  More than one race | 3 | 2 | 3 | 1 | 9
  Other | 3 | 3 | 3 | 0 | 9
  Unknown or refused to answer | 0 | 3 | 2 | 4 | 9
  Missing | 0 | 3 | 0 | 0 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5 | 2 | 12
  Not Hispanic or Latino | 86 | 51 | 109 | 55 | 301
  Unknown or Refused to Answer | 0 | 4 | 0 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 88 | 58 | 114 | 60 | 316

OUTCOME MEASURES:

1. Primary Outcome: Days of Risky Opioid Use in Past 180 Days
Description: Self-reported number of days of risky (illicit or nonmedical) opioid use in the past 180 days, assessed at 6 months after the baseline visit using single items from the Addiction Severity Index. Illicit opioid use includes use of heroin or synthetic opioids. Nonmedical opioid use includes using prescribed opioids more frequently or at higher doses than instructed on the prescription (e.g., taking 2 tablets when the prescription indicates a dose of 1 tablet), or taking pharmaceutical opioids that were not prescribed to them. Prescribed opioids may be prescribed by the participating PCP or by another medical provider. The measure is calculated as the sum of all days of use reported on the assessments of past 30-day drug use for the first 6 months (i.e., the sum of days of use from the measures collected on days 30, 60 90, 120, 150 and 180).
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 75 | 101
days | 12.2 (27.73) | 15.5 (32.64)

2. Secondary Outcome: Days of Risky Opioid Use in Past 180 Days
Description: Self-reported number of days of risky (illicit or nonmedical) opioid use in the past 180 days, assessed at 12 months after the baseline visit using single items from the Addiction Severity Index. Illicit opioid use includes use of heroin or synthetic opioids. Nonmedical opioid use includes using prescribed opioids more frequently or at higher doses than instructed on the prescription (e.g., taking 2 tablets when the prescription indicates a dose of 1 tablet), or taking pharmaceutical opioids that were not prescribed to them. Prescribed opioids may be prescribed by the participating PCP or by another medical provider. The measure is calculated as the sum of all days of use reported on the assessments of past 30-day drug use for months 7-12.
Time Frame: Month 7 up to Month 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 78 | 103
days | 10.7 (30.14) | 10.1 (27.75)

3. Secondary Outcome: Days of Benzodiazepine Use in Past 180 Days
Description: Measures of substance use are calculated as the sum of consecutive assessments of days of use in the past 30 days for the first 6 months (i.e., the sum of days of use from the measures collected on days 30, 60 90, 120, 150 and 180).
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 75 | 103
days | 2.4 (11.05) | 4 (18.66)

4. Secondary Outcome: Days of Benzodiazepine Use in Past 180 Days
Description: Measures of substance use are calculated as the sum of consecutive assessments of days of use in the past 30 days for months 7-12.
Time Frame: Month 7 up to Month 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 79 | 103
days | 2.9 (10.8) | 3 (16.36)

5. Secondary Outcome: Days of Stimulant Use in Past 180 Days
Description: as for outcome 3
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 103
days | 1.2 (8.10) | 0.6 (3.54)

6. Secondary Outcome: Days of Stimulant Use in Past 180 Days
Description: Measures of substance use are calculated as the sum of consecutive assessments of days of use in the past 30 days for months 7-12 (i.e., the sum of days of use from the measures collected on days 30, 60 90, 120, 150 and 180).
Time Frame: Month 7 up to Month 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 79 | 103
days | 2.0 (15.41) | 0.9 (4.30)

7. Secondary Outcome: Days of Marijuana Use in Past 180 Days
Description: as for outcome 3
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 75 | 103
days | 34.3 (61.47) | 31.0 (55.19)

8. Secondary Outcome: Days of Marijuana Use in Past 180 Days
Description: Measures of substance use are calculated as the sum of consecutive assessments of days of use in the past 30 days for months 7-12(i.e., the sum of days of use from the measures collected on days 30, 60 90, 120, 150 and 180).
Time Frame: Month 7 up to Month 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 79 | 103
days | 33.2 (61.19) | 34.0 (58.38)

9. Secondary Outcome: Days of Other Drug Use (Not Including Opioids, Benzodiazepines, Stimulants, and Marijuana) in Past 180 Days.
Description: as for outcome 3
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 82 | 108
days | 0.0 (0.25) | 0.1 (0.69)

10. Secondary Outcome: Days of Other Drug Use (Not Including Opioids, Benzodiazepines, Stimulants, and Marijuana) in Past 180 Days.
Description: as for outcome 6
Time Frame: Month 7 up to Month 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 82 | 108
days | 0.0 (0.11) | 0.0 (0.35)

11. Secondary Outcome: Days of Binge Alcohol Use in Past 180 Days
Description: Measures of substance use are calculated as the sum of consecutive assessments of days of use in the past 30 days for the first 6 months (i.e., the sum of days of use from the measures collected on days 30, 60 90, 120, 150 and 180). Binge alcohol use defined as 5+ drinks/day for men under age 65 and 4+ drinks/day for women and men age 65 and over.
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 76 | 103
days | 7.3 (18.06) | 9.9 (23.01)

12. Secondary Outcome: Days of Binge Alcohol Use in Past 180 Days
Description: Measures of substance use are calculated as the sum of consecutive assessments of days of use in the past 30 days for months 7-12 (i.e., the sum of days of use from the measures collected on days 30, 60 90, 120, 150 and 180). Binge alcohol use defined as 5+ drinks/day for men under age 65 and 4+ drinks/day for women and men age 65 and over.
Time Frame: Month 7 up to Month 12
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 79 | 103
days | 7.0 (21.76) | 11.2 (28.47)

13. Secondary Outcome: Number of Participants With Opioid Use Disorder
Description: Opioid use disorder is assessed using the opioid items from the modified World Mental Health Composite International Diagnostic Interview (CIDI).
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 104
Participants | 1 | 13

14. Secondary Outcome: Number of Participants With Opioid Use Disorder
Description: as for outcome 13
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 71 | 103
Participants | 3 | 6

15. Secondary Outcome: Number of Participants With Drug (Other Than Opioid) Use Disorder
Description: Drug use disorder is assessed using the drug items from the Psychiatric Diagnostic Screening Questionnaire (PDSQ).
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 101
Participants | 6 | 25

16. Secondary Outcome: Number of Participants With Drug (Other Than Opioid) Use Disorder
Description: Drug use disorder is assessed using the drug items from the Psychiatric Diagnostic Screening Questionnaire (PDSQ).
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 102
Participants | 8 | 22

17. Secondary Outcome: Number of Participants With Alcohol Use Disorder
Description: Alcohol use disorder is assessed using the alcohol items from the Psychiatric Diagnostic Screening Questionnaire (PDSQ).
Time Frame: Month 6
Measure: Count of Participants; unit: Participants
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 101
Participants | 10 | 26

18. Secondary Outcome: Number of Participants With Alcohol Use Disorder
Description: Alcohol use disorder is assessed using the alcohol items from the Psychiatric Diagnostic Screening Questionnaire (PDSQ).
Time Frame: Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 102
Participants | 9 | 20

19. Secondary Outcome: Change in Overdose Risk Behavior Questionnaire Score
Description: 13-item questionnaire assessing overdose risk behaviors. Items are rated on a Likert scale from 1 (rarely) to 4 (very often). The total score is the sum of responses and ranges from 13 to 52; higher scores indicate more prevalent overdose risk behaviors.
Time Frame: Baseline, Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 72 | 103
score on a scale | -1.43 (2.75) | -1.25 (3.03)

20. Secondary Outcome: Change in Overdose Risk Behavior Questionnaire Score
Description: as for outcome 19
Time Frame: Baseline, Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 99
score on a scale | -1.61 (3.37) | -1.15 (3.07)

21. Secondary Outcome: Episodes of Non-Fatal Overdose
Description: Number of non-fatal drug or alcohol overdoses per participant.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 103
episodes | 0.7 (5.85) | 0.7 (4.53)

22. Secondary Outcome: Episodes of Non-Fatal Overdose
Description: Number of non-fatal drug or alcohol overdoses per participant.
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: episodes
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 100
episodes | 0.3 (1.66) | 0.3 (1.11)

23. Secondary Outcome: Brief Pain Inventory (BPI) Short Form Modified Score - Pain Severity
Description: Items 3-6 from the BPI short form will be completed to assess pain severity. Items 3-6 are rated on a Likert scale from 0 (no pain) to 10 (pain as bad as you can imagine). The total score is the average of the response scores and ranges from 0-10; higher scores indicate greater pain severity.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 102
score on a scale | 4.46 (2.2) | 4.34 (2.56)

24. Secondary Outcome: Brief Pain Inventory (BPI) Short Form Modified Score - Pain Severity
Description: as for outcome 23
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 102
score on a scale | 4.46 (2.29) | 3.98 (2.58)

25. Secondary Outcome: Brief Pain Inventory (BPI) Short Form Modified Score - Pain Interference
Description: Items 9A-9G from the BPI short form will be completed to assess pain interference. Items 9A-9G are rated on a Likert scale from 0 (does not interfere) to 10 (completely interferes). The total score is the average of the response scores and ranges from 0-10; higher scores indicate greater pain interference.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 102
score on a scale | 4.38 (2.91) | 4.32 (2.87)

26. Secondary Outcome: Brief Pain Inventory (BPI) Short Form Modified Score - Pain Interference
Description: as for outcome 25
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 102
score on a scale | 4.14 (2.79) | 3.87 (2.8)

27. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Anxiety Short Form Score
Description: The PROMIS Anxiety Short Form comprises 8 questions assessing anxiety. Each item is rated on a scale from 1 (never) to 5 (always). The raw score is the sum of responses and ranges from 8 to 40. The raw score is converted to a standardized t-score ranging from 0-100 with a mean of 50 and a standard deviation of 10. Higher t-scores indicate greater levels of anxiety.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 102
T-score | 9.99 (8.59) | 9.66 (7.78)

28. Secondary Outcome: PROMIS Anxiety Short Form Score
Description: as for outcome 27
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 102
T-score | 10.27 (8.91) | 9.63 (7.83)

29. Secondary Outcome: Patient Health Questionnaire-8 (PHQ-8) Score
Description: The Patient Health Questionnaire-8 (PHQ-8) is a self-reported questionnaire that measures depressive symptoms. The PHQ-8 score is calculated by adding up the scores from each of the eight items on the questionnaire. The score ranges from 0 to 24, with higher scores indicating more severe depression.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 104
score on a scale | 5.77 (5.16) | 6.53 (5.63)

30. Secondary Outcome: Patient Health Questionnaire-8 (PHQ-8) Score
Description: as for outcome 29
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 72 | 102
score on a scale | 6.39 (5.69) | 5.68 (4.68)

31. Secondary Outcome: Health-Related Quality of Life (SF-12) - Physical Component Summary (PCS)
Description: Health-Related Quality of Life (SF-12) is a 12-item assessment of quality of life. The Physical Component Summary (PCS) subscale comprises physical health-related questions in the SF-12. The PCS raw score is the sum of responses. The PCS raw score is converted into a total score ranging from 0-100; higher scores indicate better physical health.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 103
score on a scale | 39.43 (10.63) | 40.45 (11.48)

32. Secondary Outcome: Health-Related Quality of Life (SF-12) - Physical Component Summary (PCS)
Description: as for outcome 31
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 102
score on a scale | 39.51 (10.99) | 41.84 (11.84)

33. Secondary Outcome: Health-Related Quality of Life (SF-12) - Mental Component Summary (MCS)
Description: Health-Related Quality of Life (SF-12) is a 12-item assessment of quality of life. The Mental Component Summary (MCS) subscale comprises mental health-related questions in the SF-12. The MCS raw score is the sum of responses. The MCS raw score is converted into a total score ranging from 0-100; higher scores indicate better mental health.
Time Frame: Month 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 103
score on a scale | 46.56 (12.32) | 47.01 (11.26)

34. Secondary Outcome: Health-Related Quality of Life (SF-12) - Mental Component Summary (MCS)
Description: as for outcome 33
Time Frame: Month 12
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 102
score on a scale | 46.11 (11.59) | 46.05 (9.32)

35. Secondary Outcome: Number of Acute Care Events
Description: Measured as the total number of self-reported emergency department (ED) visits in the past six months.
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 103
Events | 0.37 (0.76) | 0.36 (0.81)

36. Secondary Outcome: Number of Acute Care Events
Description: Measured as the total number of self-reported emergency department (ED) visits in the past six months.
Time Frame: Month 7 up to Month 12
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 100
Events | 0.45 (0.76) | 0.30 (0.73)

37. Secondary Outcome: Number of Acute Care Events (Self-Report)
Description: Measured as the total number of self-reported hospital utilizations in the past six months.
Time Frame: Up to Month 6
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 73 | 103
Events | 0.26 (0.91) | 0.12 (0.38)

38. Secondary Outcome: Number of Acute Care Events (Self-Report)
Description: Measured as the total number of self-reported hospital utilizations in the past six months.
Time Frame: Month 7 up to Month 12
Measure: Mean (Standard Deviation); unit: Events
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 74 | 100
Events | 0.28 (0.96) | 0.20 (0.92)

ADVERSE EVENTS:
Time Frame: Serious and Other [Not Including Serious] Adverse Events were not monitored/assessed among patient participants nor PCPs. All-cause mortality was assessed among patient participants, but not among PCPs.
Description: 12 months
Arm/Group | Subthreshold Opioid Use Disorder Prevention(STOP) Intervention | Enhanced Usual Care (EUC)
All-Cause Mortality (participants affected / at risk) | 0/88 | 2/114
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT04218201/Prot_002.pdf
  • Statistical Analysis Plan (2025-05-23): https://cdn.clinicaltrials.gov/large-docs/01/NCT04218201/SAP_003.pdf
  • Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT04218201/ICF_000.pdf